CLINICAL TRIAL: NCT02321644
Title: A Two-Part, Phase 1 Study to Evaluate Pharmacokinetics and Pharmacodynamics of Multiple Dose CC-90001 and to Evaluate the Effects of Food and Formulation on Pharmacokinetics of Single Dose CC-90001 in Healthy Subjects
Brief Title: Effect of UV Exposure on the PD of Multiple Doses of CC-90001 and Pilot Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90001-CP-002
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Subjects
Keywords: CC-90001; PHARMACOKINETICS; PHARMACODYNAMICS; HEALTHY SUBJECTS; SINGLE DOSE; MULTIPLE DOSE; PUNCH BIOPSY
MeSH Terms: interventions — CC-90001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CC-90001 (Experimental): Part 1: All subjects will receive the following doses of CC-90001 in the fixed sequence below:
  Treatment A: 60 mg CC-90001 as Active-Ingredient-in-Capsule, once daily x 6 days Treatment B: 160 mg CC-90001 as Active-Ingredient-in-Capsule, once daily x 6 days Treatment C: 400 mg of CC-90001 as Active-Ingredient-in-Capsule, once daily x 6 days
  Interventions: Drug: CC-90001
- CC-90001 2 X 100mg fasted (Experimental): Treatment D: 2 x 100 mg CC-90001 as Active-Ingredient-in-Capsule, single oral dose administered under fasted conditions.
  Interventions: Drug: CC-90001
- CC-90001 1 X 200mg fasted (Experimental): Treatment E: 1 x 200 mg CC-90001 [formulated tablet(s)] single oral dose administered under fasted conditions
  Interventions: Drug: CC-90001
- CC-90001 1 X 200mg fed (Experimental): Treatment F: 1 x 200 mg CC-90001 [formulated tablet(s)] single oral dose administered under fed conditions (standard high fat breakfast).
  Interventions: Drug: CC-90001

INTERVENTIONS:
Drug: CC-90001 — CC-90001 Active-ingredient-in-capsule and formulated tablet

SUMMARY:
This is a two-part, phase 1 study to evaluate the pharmacokinetics and pharmacodynamics of multiple doses of CC-90001 and the effects of food and formulation on the pharmacokinetics of single dose CC-90001 in healthy subjects. Part 1 involves the exposure of subjects to the minimum amount of UV-B light that causes minimally perceptible skin reddening. This will take place before dosing (baseline) and 3 times more while on increasing doses of CC-90001. Punch biopsies of the exposed areas will be taken and assessed for c-Jun terminal kinase activity. Part 2 involves evaluation of changes in pharmacokinetics of 2 formulations of CC-90001 when administered in the fasted state and after a high-fat meal.

DETAILED DESCRIPTION:
Part 1 is an open-label, multiple-dose, 3-period, fixed-sequence study, to evaluate the effect of CC-90001 on JNK activity following UV irradiation. On the first day prior to dosing (baseline), and on the 6th day of each dosing period (Days 6, 12, and 18), twice the MED intensity of UV light will be administered to delineated sites on the subjects' buttocks. The irradiation at baseline (Day -1) should be administered at approximately the same time that irradiation is scheduled on Days 6, 12, and 18, which is at 2 hours post dose. Eight hours after UV irradiation, a skin punch biopsy will be taken from the UV exposure site. The end of confinement will be Day 19. The follow-up visit will occur 7-10 days (ie, Day 25 to Day 28) following the last dose in Period 3. An early termination (ET) visit will occur within 10 days of the day of discontinuation. The MED will be determined within 10 days of dosing in Period 1. All subjects will receive the following doses of CC-90001 in the fixed sequence below: Treatment A: 60 mg CC-90001 as AIC, QD x 6 days; Treatment B: 160 mg CC-90001 as AIC, QD x 6 days; and Treatment C: 400 mg of CC-90001 as AIC, QD x 6 days. Subjects will be confined at the unit from Day -1 until discharge on Day 19 after all safety assessments.

In Part 2 subjects will be assigned randomly to one of three dosing sequences during which they will receive one of the following dosing regimens:

* Treatment D: 2 x 100 mg CC-90001 as AIC, single oral dose administered under fasted conditions.
* Treatment E: 1 x 200 mg CC-90001 [formulated tablet(s)] single oral dose administered under fasted conditions
* Treatment F: 1 x 200 mg CC-90001 [formulated tablet(s)] single oral dose administered under fed conditions (standard high fat breakfast).

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign a written Informed Consent Document (ICD) prior to any study-related assessments/procedures being performed
2. Must be able to communicate with the Investigator and to understand and adhere to the study visit schedule and other protocol requirements
3. Must be a male or female*, aged 18 years of age to 65 years of age (inclusive) at the time of signing the ICD

   * Women of child-bearing potential (WCBP)*must agree to ongoing pregnancy testing during the course of the study, and at the end of the study. This applies even if the subject practices true abstinence from heterosexual contact
   1. The female subjects must either commit to true abstinence** from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, 2 highly effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including dose interruptions), and for at least 28 days after discontinuation of study drug
   2. Females not of child-bearing potential should have been either surgically sterilized at least 6 months prior to screening (hysterectomy or bilateral tubal ligation) or be postmenopausal (defined as 24 months with no menses prior to Screening, AND with a plasma follicle stimulating hormone (FSH) > 40 IU/L at screening). Documentation will be required in cases of tubal ligation
4. Males must practice true abstinence** or agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a WCBP while on study drug, or while participating in this study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy

   ** True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception]
5. Has a body mass index (BMI = weight [kg]/(height [m2]) between 18 and 33 kg/m2 (inclusive)
6. Must be healthy as determined by the Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECGs

   * Must be afebrile (febrile is defined as ≥ 38 °C or 100.3° Fahrenheit)
   * Systolic blood pressure must be in the range of 80 to 140 mmHg, diastolic blood pressure must be in the range of 40 to 90 mmHg, and pulse rate must be in the range of 40 to 110 bpm
   * QTcF value ≤ 430 msec for male subjects and ≤ 450 msec for female subjects. An ECG may be repeated up to 3 times to determine subject eligibility
7. Additional criteria for Part 1 only:

   1. Must be Fitzpatrick skin type I or II
   2. Must have a valid MED obtained within 10 days prior to dosing

Exclusion Criteria:

1. History (ie, within 3 years) of any clinically significant neurological, gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other major disorders
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study, or confounds the ability to interpret data from the study
3. Use of any prescribed systemic or topical medication, including vaccines, within 30 days of the first dose
4. Use of any non-prescribed systemic or topical medication (including herbal medicines) within 14 days of the first dose administration (with the exception of vitamin/mineral supplements)
5. Use of any metabolic enzyme inhibitors or inducers (ie, CYP3A inducers and inhibitors or St. John's wort) within 30 days of the first dose administration

   a. The University of Indiana "Cytochrome P450 Drug Interaction Table" should be used to determine inhibitors and/or inducers of CYP 3A4 (http://medicine.iupui.edu/clinpharm/ddis/table/aspx)
6. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME), eg, bariatric procedure

   a. Appendectomy and cholecystectomy are acceptable
7. Donated blood or plasma within 8 weeks before the first dose administration
8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs)
9. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or positive alcohol screen
10. Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb), or have a positive result to the test for HIV antibodies at Screening
11. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer)
12. Smoke more than 10 cigarettes per day, or the equivalent in other tobacco products (self reported)
13. Subject has a history of multiple drug allergies (ie, 2 or more)

Additional Exclusion Criteria for Subjects in Part 1 Only:

1. Inability to evaluate the skin in and around the test sites due to sunburn, tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or any other disfiguration
2. Used any creams or lotions (ie, containing sun protection factor [SPF]) in the test area (ie, buttocks) within 7 days of study start (Day 1)
3. Participation in any test for irritation or sensitization or any test involving UV exposures on the test area within four weeks of study start
4. Participation in another study requiring biopsy (on the planned test area) within the past 2 months
5. History of wound healing or blood-clotting abnormality
6. History of keloid formation or hypertrophic scarring following skin injury
7. History of severe reactions from exposure to sunlight
8. History of allergy to lidocaine or other similar local anesthetics
9. History of allergy to epinephrine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics- Cmax | Days 1, 2, 3, and 4
  Maximum observed plasma concentration
Pharmacokinetics- Tmax | Days 1, 2, 3, and 4
  Time to Cmax
Pharmacokinetics- AUC∞ | Days 1, 2, 3, and 4
  Area under the plasma concentration time curve from time zero extrapolated to infinity
Pharmacokinetics- AUCt | Days 1, 2, 3, and 4
  Area under the plasma concentration time curve from time zero to the last quantifiable concentration
Pharmacokinetics- AUCτ | Days 1, 2, 3, and 4
  Area under the plasma concentration-time curve from time zero to tau, where tau is the dosing interval
Pharmacokinetics- t1/2 | Days 1, 2, 3, and 4
  Terminal phase elimination half-life
Pharmacokinetics- CL/F | Days 1, 2, 3, and 4
  Apparent total plasma clearance when dosed orally
Pharmacokinetics- Vz/F | Days 1, 2, 3, and 4
  Apparent total volume of distribution when dosed orally, based on the terminal phase
Pharmacodynamics: Phospho-c-Jun IHC data will be subjectively scored on a scale of 0 to 4 based on the intensity and number of epidermal keratinocyte nuclei stained within the tissue section by trained individuals blinded to treatment | Approximately 6 days
  For Part 1 only the Phospho-c-Jun IHC data will be subjectively scored on a scale of 0 to 4 based on the intensity and number of epidermal keratinocyte nuclei stained within the tissue section by trained individuals blinded to treatment.

SECONDARY OUTCOMES:
Adverse Event (AE) | approximately 10 weeks
  An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. AE will be monitored, evaluated, recorded and reported by using following:
  * Physical examinations (PEs)
  * Vital sign measurements
  * 12 lead electrocardiograms (ECGs)
  * Clinical laboratory safety tests
  * Concomitant medications and procedures

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Study Director — Celgene Corporation
Locations (2):
- United States (2):
  - Covance-Daytona Beach, Daytona Beach, Florida
  - TKL Research, Fair Lawn, New Jersey